CLINICAL TRIAL: NCT04290754
Title: PATH 2 Purpose: Primary Care and Community-Based Prevention of Mental Disorders in Adolescents
Acronym: P2P
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Illinois College of Medicine Rockford (Other); Wake Forest University Health Sciences (Other); Katherine Shaw Bethea Hospital (Unknown); University of Louisville (Other); Patient-Centered Outcomes Research Institute (Other); Brown University (Other); Mile Square Health Center (Other)
Responsible Party: Principal Investigator, Benjamin Van Voorhees, MD, MPH, Professor of Medicine, Head of Department of Pediatrics, Physician-in-Chief of Childrens Hospital University of Illinois, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CHAIRb 19081501; IHS-2017C3-9333 (Other Grant/Funding Number: PCORI); 094637 (Other: UIC ORS Award Number)
Record Dates: First submitted 2020-02-10; First posted 2020-03-02 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-12

CONDITIONS: Depression
Keywords: Adolescents; Depression; Internet intervention; Cognitive-Behavioral Therapy; Prevention; Group Therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Comparative Effectiveness Study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Cluster randomization of clinic sites
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CATCH-IT (Experimental): Competent Adulthood Transition with Cognitive-behavioral & Interpersonal Training (CATCH-IT) is an internet-based depression prevention program that targets decreasing modifiable risk factors while enhancing protective factors in at-risk adolescents, and that includes a parent program. It has been shown to be safe, feasible, and efficacious.
  Interventions: Behavioral: CATCH-IT
- TEAMS (Active Comparator): Teens Achieving Mastery over Stress (TEAMS) is an 8-session group depression prevention program teaching teens how to deal with stress and negative moods, and ways to manage low mood based on cognitive-behavioral therapy (CBT) principles and strategies. Efficacy has been demonstrated by several trials over time.
  Interventions: Behavioral: TEAMS

INTERVENTIONS:
Behavioral: CATCH-IT — Competent Adulthood Transition with Cognitive-behavioral & Interpersonal Training (CATCH-IT) is an internet-based depression prevention program that targets decreasing modifiable risk factors while enhancing protective factors in at-risk adolescents, and that includes a parent program. It has been shown to be safe, feasible, and efficacious.
  Arms: CATCH-IT
Behavioral: TEAMS — Teens Achieving Mastery over Stress (TEAMS) is an 8-session group depression prevention program teaching teens how to deal with stress and negative moods, and ways to manage low mood based on cognitive behavioral therapy (CBT) principles and strategies. Efficacy has been demonstrated by several trials over time.
  Other Names: Prevention of Depression (POD)
  Arms: TEAMS

SUMMARY:
PATH (Promoting AdolescenT Health) 2 Purpose is a two-arm comparative effectiveness research trial to that will evaluate the ability of the interventions, Competent Adulthood Transition with Cognitive-behavioral & Interpersonal Training (CATCH-IT) and Teens Achieving Mastery over Stress (TEAMS), to intervene early to prevent depressive illness and potentially other common mental health disorders. Using cluster randomization, 564 participants eligible for the study will be offered one of two different depression prevention programs in multiple sites in Chicagoland, Rockford, Illinois; Dixon, Illinois; and Louisville, Kentucky. In response to the Coronavirus Disease 2019 (COVID-19) pandemic, we will employ a public health media campaign to recruit a second cohort of 100 adolescents state-wide in Illinois, Kentucky, and Massachusetts individually randomized to either intervention. The study will also assess teens', parents' and providers' experiences with each intervention approach. Finally, we will examine the impact of the COVID-19 pandemic on adolescents at-risk for depression who are enrolled in our study.

DETAILED DESCRIPTION:
The majority of mental, emotional and behavioral (MEB) disorders have an initial onset before age 24, with 20% annual incidence, with major depressive disorder (MDD) being the most common MEB. Health systems, eager to reduce costs, want to transition from the current "wait until sick enough for treatment" model for MDD to a preventive model. However, evidence is needed for (1) the comparative effectiveness of a "scalable intervention" and (2) an implementation model for such a scalable intervention in the primary care setting. This study is a comparative effectiveness trial evaluating the efficacy of two evidence-based cognitive-behavioral prevention (CBP) programs: Teens Achieving Mastery over Stress (TEAMS), the "gold standard," group therapy model, and Competent Adulthood Transition with Cognitive Behavioral, Humanistic and Interpersonal Training (CATCH-IT), a scalable, self-directed, technology-based model. For implementation during the COVID-19 pandemic, TEAMS has successfully been adapted to an online format and administered online through HIPAA-compliant video conferencing software. For the first cohort, 564 eligible adolescents age 13-18 will be offered one of two different depression prevention programs using cluster randomization in multiple sites in urban and suburban Chicago, Illinois; rural Western Illinois, including Dixon and surrounding towns; and Louisville, Kentucky. Randomization will be blocked into matched pairs of primary health care clinics and school sites and stratified by race, ethnicity, rural-urban commuting area codes, and socio-economic disadvantage using the Distressed Communities Index (DCI) from census-tracked data of each site zip code. A second cohort of 100 eligible adolescents will be recruited through public health media campaigns in Illinois, Kentucky, and Massachusetts utilizing the same eligibility criteria as Cohort One. These participants will connect with the research team by phone, email, web survey, or social media and will be randomized at the individual-level with equal allocation into treatment conditions (CATCH-IT or TEAMS). The investigators will comprehensively evaluate patient-centered outcomes and stakeholder-valued moderators of effect at 2, 6, 12, and 18 month assessment points. Using a hybrid clinical trial design that simultaneously examines implementation process, the study will also assess adolescents', parents' and providers' experiences (i.e. efficacy, time commitment, cultural acceptability, and implementation cost) with each intervention approach. A sub-sample of Cohort Two (n=50, 25 from each intervention arm) will be recruited to participate in open-ended interviews for adolescents to share their experiences of living with subsyndromal depression, coping during the COVID-19 pandemic, their perceived impact of CATCH-IT or TEAMS on their mood and behavior, and the cultural contexts in which these experiences occurred.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 13 through 19 years, and
* Adolescent must be experiencing an elevated level of depressive symptoms (Patient Health Questionnaire-9 Score = 5-18), and
* Adolescent will be included if they have a past, but not current history of depression.

Exclusion Criteria:

* Outside age range
* A current diagnosis of Major Depression
* Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) diagnosis of: schizophrenia, bipolar affective disorder, extreme current drug or alcohol abuse.
* Currently using medication therapy for depression, anxiety, or other internalizing disorders for less than 3 months.
* Currently engaged in individual treatment for a mood disorder
* Currently engaged in a cognitive-behavioral group or therapy
* Any past psychiatric hospitalizations
* Any past self-harm attempt with moderate or greater lethality
* Current suicidal thoughts
* Not willing to comply with the study protocol
* Not willing to participate in the TEAMS groups
* Not willing to be audio recorded during TEAMS groups (only for TEAMS clinics)
* Unable to complete the PHQ-9 screening due to cognitive or intellectual impairment
* Did not complete phone assessment with MINI Kid
* Parent/guardian has a cognitive or intellectual impairment.
* Participant Declined/Changed Mind/Uninterested in participating

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 636 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Time | Baseline through 18 months
  Time will be measured to nearest minute for all intervention related activities including initial screening, engagement phone calls, use of CATCH-IT, TEAMS group activities, including travel time to and from TEAMS groups. Time will be measured from adolescent, family, practice, community center, healthcare organization, health system perspective. For time that cannot be directly measured by study staff, the investigators will sample direct observation or questionnaires to capture time required for health system related activities such as screening and engagement.
Cultural acceptability adolescent and family | Baseline through 18 months
  Cultural acceptability for each stakeholder using appropriate, validated instruments. Adolescent and family: Usefulness, Satisfaction, and Ease Questionnaire (USE, 30 items, self-report, 7-point Likert scale, 30-210 score range, higher score indicates more acceptable). An example statement is: "I would recommend this to a friend."
Cost | Baseline through 18 months
  Costs will be measured for all stakeholders. For practice, community center, healthcare organizations, health systems, cost will be measured to nearest dollar by converting time measures into employment related costs based on mean wages an benefits for staff at that occupational level. Adolescent and family costs will be measured by converting time into mean hourly wages and benefits for adolescent and family members involved in the project (based on mean wage for age and occupation).
Depressive and mental disorder episodes | Baseline through 18 months
  Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI Kid, self-report). This is a structured psychiatric interview administered by a trained staff member which uses stem questions and follow-ups to determine the presence of symptoms and date of onset. The staff member then determines if and when the symptoms developed an episode is present. Measure is either episode present or not and date of onset.
Stress symptoms | Baseline through 18 months
  Center for Epidemiological Studies-Depression Scale (CES-D, 20 items, self-report, measured in frequency, 0,"not at all" to 3, "nearly every day in last week, 0-60 score range, higher score indicates more depressed)
Resiliency | Baseline through 18 months
  Resiliency will be measured across multiple domains. To assess resiliency in terms of coping skills, the Connor-Davidson Resilience Scale (CD-RISC, 10 items, self-report, 4 levels of response, 0-40 score range, higher score indicates better coping skills)
Function | Baseline through 18 months
  Social Adjustment Scale Self-Report (SAS-SR, 23-items, self-report, 5-point Likert scale, 23-115 score range, higher score indicates higher levels of social adjustment) administered to adolescents only.
Relationships (Life Events) | Baseline through 18 months
  University of California at Los Angeles (UCLA) Life Events Scale (19-items, self-report) administered to adolescents only.
Socio-cultural Relevance | Baseline through 18 months
  The Socio-Cultural Relevance Scale (10-item and 14-item versions, self-report, 5-point Likert scale, 10-40 or 14-56 score ranges, higher score indicates greater socio-cultural relevance) will assess perceived change and satisfaction with the intervention, component of cultural acceptability to adolescent)
Organizational Readiness to Change Assessment | Baseline
  Organizational Readiness to Change Assessment (ORCA, 18 questions, 4 items per question, self-report, 5-point Likert scale, 18-90 score range, higher score indicates higher organizational readiness, component of cultural acceptability to practice, community center, healthcare organizations, health systems)
Intervention Sustainability | end of study, 30 months
  Program Sustainability Assessment Tool (PSAT, 8 questions, self-report 5 items per question, 7-point Likert scale, 8-56 score range, higher score indicates higher capacity for program sustainability, component of cultural acceptability to practice, community center, healthcare organizations, health systems)
Acceptability of Intervention | end of study, 30 months
  Acceptability of Intervention Measure (AIM, 1 question with 4 items, self-report, 5-point Likert scale, 1-5 score range, higher score indicates greater acceptability of intervention, to be completed by all staff and leadership, repeatedly, component of cultural acceptability to practice, community center, healthcare organizations, health systems)
Feasibility of Intervention | end of study, 30 months
  Feasibility of Intervention Measure (FIM, 1 question with 4 items, self-report, 5-point Likert scale, 1-5 score range, higher score indicates greater feasibility of intervention, to be completed by all staff and leadership, repeatedly, component of cultural acceptability to practice, community center, healthcare organizations, health systems)
Intervention Appropriateness | Baseline through 18 months
  Intervention Appropriateness Measure (IAM, 1 question with 4 items, self-report, 5-point Likert scale, 1-5 score range, higher score indicates greater appropriateness of intervention, to be completed by all staff and leadership, repeatedly, component of cultural acceptability to practice, community center, healthcare organizations, health systems)
Depressive Symptoms | Baseline through 18 months
  Patient Health Questionnaire-Adolescent (PHQ-A, 9 items plus 4 follow-up items, self-report, 3-point Likert scale, 0-27 score range, higher score indicates more depression symptoms/severity)
Externalizing Behavior Symptoms | Baseline through 18 months
  Disruptive Behavior Disorders Rating Scale-Adolescent (DBD-A, 41-items, self-report, 4-point Likert scale, 0-123 score range, higher score indicates greater externalizing symptoms)
Anxiety Symptoms | Baseline through 18 months
  Screen for Child Anxiety Related Disorders (SCARED, 41-items, self-report, 3-point Likert scale, 0-82 score range, higher score indicates greater anxiety symptoms)
Substance Abuse Symptoms | Baseline through 18 months
  Car, Relax, Alone, Forget, Friends, Trouble substance use assessment (CRAFFT, 6 items, self-report, 2-point scale, 0-6 score range, higher score indicates greater substance abuse symptoms)
Post Traumatic Stress Disorder Symptoms | Baseline through 18 months
  Child Post Traumatic Symptoms Disorder Scale (24-items, self-report, 4-point Likert scale, 0-72 score range, higher score indicates greater PTSD symptom levels)
Rumination | Baseline through 18 months
  Tendency towards rumination will be assessed by the Children's Response Style Scale (CRSS, 10-items, self-report, 5-point Likert scale, 0-50 score range, higher score indicates greater rumination (more repeated negative thinking, less resilient, component of resiliency)
Dysfunctional Attitudes | Baseline through 18 months
  The Dysfunctional Attitude Scale (DAS, 9-item, self-report, 7-point Likert scale, 9-63 score range, higher score indicates more dysfunctional attitude, less resiliency, component of resiliency)
Relationships-Family | Baseline through 18 months
  Child Report of Parental Behavior Inventory (CRPBI, 30-item, self-report, 3-point Likert scale, 0-60 score range, higher scores indicate more positive parent child relationship).
Blood Pressure | Baseline and 18 months
  Measured in millimeters of mercury
Body Mass Index | Baseline and 18 months
  Calculated by measuring height (centimeters) and weight (kilogram) to calculate kg/meters squared (BMI, Body Mass Index)
Weight | Baseline and 18 months
  Measured in kilograms by standard medical office scale, fully clothed participant
Height | Baseline and 18 months
  Measure by standard medical office practice measure, without shoes, in centimeters
Recruiting model and comparative effectiveness outcomes | Baseline through 18 months
  With the addition of a second cohort to be recruited through a public health media campaign, we will compare results between groups in each arm, and between the two recruitment models. We will compare implementation and clinical outcomes in the same trial arm, but also across the two recruiting methods.

SECONDARY OUTCOMES:
Implementation themes | End of study, 30 months
  Consolidated Framework for Implementation Research (CFIR) will be used to explore experience of the study from the perspective of 25 stakeholders
Moderation of Covid-19 factors on comparative effectiveness outcomes | Baseline through 18 months
  We will examine factors related to the COVID-19 pandemic that may be moderators of study outcomes: (1) COVID-19-related behaviors and consequences (e.g. social distancing, sheltering-in-place, family illness and death), and (2) Social determinants of health (e.g. food insecurity, internet access, unemployment) in both cohorts using the Holliston at-Home Questionnaire (a 26-item, adolescent self-report, 5-point Likert scale, 0-150 score range, higher score indicates greater externalizing symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Van Voorhees, MD, MPH, Principal Investigator — University of Illinois at Chicago, School of Medicine; Tracy RG Gladstone, PhD, Principal Investigator — Wellesley College, Wellesley Centers for Women
Locations (1):
- UI Health, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knepper AK, Feinstein RT, Sanchez-Flack J, Fitzgibbon M, Lefaiver C, McHugh A, Gladstone TRG, Van Voorhees BW. Primary care-based screening and recruitment for an adolescent depression prevention trial: Contextual considerations during a youth mental health crisis. Implement Res Pract. 2024 Apr 22;5:26334895241246203. doi: 10.1177/26334895241246203. eCollection 2024 Jan-Dec. PMID 38655380
- See also: Path2Purpose Website — https://www.path2purpose.info/